CLINICAL TRIAL: NCT07364422
Title: A Multicenter, Open-label, Single-arm, Dose-finding and Expansion Phase 1b/2 Study to Evaluate the Safety and Tolerability of JPI-547 in Combination With Irinotecan as a Third Line and Beyond Therapy for Recurrent or Metastatic Gastric Cancer
Brief Title: To Evaluate the Safety and Tolerability of Study Drug as a Third-line and Beyond Therapy for Recurrent or Metastatic Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JPI-547-103
Record Dates: First submitted 2026-01-11; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer (GC)
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JPI-547 and Irinotecan (Experimental): coadministration of JPI-547 and Irinotecan
  Interventions: Drug: JPI-547; Drug: Irinotecan (drug)

INTERVENTIONS:
Drug: JPI-547 — The dose levels will be escalated following a 3+3 dose escalation scheme.
Drug: Irinotecan (drug) — The dose levels will be escalated following a 3+3 dose escalation scheme.

SUMMARY:
This study aims to evaluate the safety and tolerability of JPI-547 in combination with irinotecan as a third-line and beyond therapy for recurrent or metastatic gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma who have progressed after second-line therapy.
* Those with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Those with at least one measurable lesion in accordance with RECIST 1.1

Exclusion Criteria:

* Patients with a confirmed specific medical history or past surgical history
* Patients who meet specific criteria regarding prior treatment
* Patients with a history of specific drug administration
* Patients with specific comorbidities.
* Patients who have undergone major surgery within 4 weeks prior to screening or are expected to require major surgery during the clinical trial are excluded. (However, those who have had minor surgeries
* Patients with symptoms at the time of screening, who have not received treatment, or who have rapidly progressing central nervous system (CNS) metastases.
* Patients with mental disorders or altered mental status/consciousness (AMS) that impair their ability to understand this clinical trial for informed consent.
* Pregnant or Lactating Women
* Subjects with a history of severe allergic anaphylactic reactions to the investigational product and/or its components, or who have contraindications to the administration of the investigational product and/or irinotecan
* Patients considered unsuitable for this clinical trial by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
1b: dose-limiting toxicity rate | The dose-limiting toxicity evaluation window is 28 days from C1D1.
phase 2: Overall Response Rate (ORR) according to RECIST v1.1 | At 6-week intervals through study completion, an average of 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, South Korea